CLINICAL TRIAL: NCT01428115
Title: Reveal the Level of Anxiety in Patients With Crohn's Disease Receiving Adalimumab
Acronym: RELAX
Status: Completed | Type: Observational
Sponsor: AbbVie (prior sponsor, Abbott) (Industry)
Collaborators: Raffeiner GmbH (Industry)
Responsible Party: Sponsor
Organization: AbbVie (Industry)
Other Study IDs: P12-705
Record Dates: First submitted 2011-09-01; First posted 2011-09-02 (Estimated); Results first posted 2014-11-03 (Estimated); Last update posted 2014-11-03 (Estimated); Status verified 2014-10

CONDITIONS: Severe Crohn's Disease; Anxiety
Keywords: monoclonal; anxiety; antibodies; adalimumab; severe crohn's disease; quality of life; biological products
MeSH Terms: conditions — Crohn Disease; Anxiety Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with severe active Crohn's disease: Patients with severe active Crohn's disease for whom adalimumab was prescribed in the usual manner in accordance with the terms of the local marketing authorization.

SUMMARY:
It has been shown that emotional health issues, such as state anxiety, are more prevalent in patients suffering from inflammatory bowel disease (IBD) compared to physically healthy subjects.

Such findings have to be taken into consideration when making an educated guess that psychological factors such as depression and anxiety in particular interact with the course of Crohns disease. Therefore the treatment of the underlying disease may have a significant influence on the level of psychological disorders.

Several studies have shown that treatment with tumor necrosis factor alpha (TNF-α) antibodies ameliorates the emotional/psychological status of patients, however the impact of adalimumab therapy on anxiety correlated with the status of inflammatory bowel disease (IBD) remains unclear.

The primary objective of this study was to describe and evaluate changes in levels of anxiety assessed by validated patient questionnaires after 6 months of treatment with adalimumab.

ELIGIBILITY:
Inclusion Criteria:

* Patients for whom Adalimumab (Humira) therapy is indicated and has been prescribed according to the product label and who meet the following criteria:

  * Male and female patients aged 18 to 65 years suffering from severe active Crohns Disease, attending a routine medical visit.
  * Able to complete questionnaires.
  * Patients with status active severe Crohns disease which required immunosuppressive treatment
  * Patients must fulfil international and national guidelines for the use of a biologic therapies in Crohns Disease (Chest X-ray and interferon gamma release assay (IGRA) or PPD (purified protein derivative)-skin test negative for tuberculosis).
  * Patients have not responded despite a full and adequate course of therapy with a corticosteroid and/or an immunosuppressant; or who are intolerant to or have medical contraindications for such therapies.
  * Patients who have been prescribed in line with the European Summary of Product Characteristics (SMPC)

Exclusion Criteria:

* The following patients will not be included in this observational study:

  * Previous therapy with TNF-α blocker within the last 8 weeks
  * Active Central Nervous System opportunistic infections or Central Nervous System malignancies.
  * History of Cerebrovascular Accident
  * Abuse of illicit substances (such as psychoactive drugs) within the previous 3 months
  * Change of medication-based treatment of generalized anxiety and panic disorder, psychiatric disorder
  * No informed consent
  * Contraindication to adalimumab (Humira) therapy according to the SMPC
  * Current or planned pregnancy
  * Lactation according to SMPC
  * Planned change of site within the next 24 weeks.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The investigational sites were centers with a high level of experience in the treatment of Crohns disease patients.
Sampling Method: Non-Probability Sample
Enrollment: 83 (Actual)
Dates: Start 2011-12; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Astrid Dworan-Timler, MD, Study Director — AbbVie Austria
Locations (8):
- Austria (8):
  - Site Reference ID/Investigator# 64830, Graz
  - Site Reference ID/Investigator# 64832, Innsbruck
  - Site Reference ID/Investigator# 64829, Linz
  - Site Reference ID/Investigator# 79613, Saint Veit/Glan
  - Site Reference ID/Investigator# 64831, Salzburg
  - Site Reference ID/Investigator# 64828, Sankt Pölten
  - Site Reference ID/Investigator# 47342, Vienna
  - Site Reference ID/Investigator# 64833, Vienna

REFERENCES:
- See also: Related Info — http://rxabbvie.com

RESULTS

PARTICIPANT FLOW:
Groups:
- Adalimumab: Participants received 40 mg every other week via subcutaneous injection according to Summary of Product Characteristics (SmPC)
Period: Overall Study
Arm/Group | Adalimumab
Started | 83
Completed | 62
Not Completed | 21
Not completed — Lack of Efficacy | 3
Not completed — Lost to Follow-up | 10
Not completed — Pregnancy | 1
Not completed — Protocol Violation | 3
Not completed — Withdrawal by Subject | 4

BASELINE CHARACTERISTICS:
Arm/Group | Adalimumab
Number analyzed (Participants) | 83
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.6 (11.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43
  Male | 40
Participants with Comorbidities [Number; unit: participants]
  Yes | 18
  No | 65

OUTCOME MEASURES:

1. Primary Outcome: Change in State Trait Anxiety Index (STAI) State Scores From Baseline to After 6 Months of Treatment With Adalimumab
Description: The STAI questionnaire consists of 40 questions with 20 items allocated to each of the State Anxiety and Trait Anxiety subscales. The scores for each subtest range from 20 to 80, with higher scores indicating higher levels of anxiety.
Time Frame: Baseline and Visit 3 [Month 6]
Population: All data were analyzed as observed and missing values were not replaced by any imputation method. In analyses of changes between visits, only patients with values at both visits were include.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Adalimumab
Number analyzed (Participants) | 59
scores on a scale | -1.7 (9.8)

2. Primary Outcome: Change in State Trait Anxiety Index (STAI) Trait Scores From Baseline to After 6 Months of Treatment With Adalimumab
Description: as for outcome 1
Time Frame: Baseline and Visit 3 [Month 6]
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Adalimumab
Number analyzed (Participants) | 57
scores on a scale | -9.0 (9.2)

3. Primary Outcome: Change in Hospital Anxiety and Depression Score (HADS) - Anxiety, From Baseline to After 6 Months of Treatment With Adalimumab
Description: HADS is used to detect emotional disturbances (such as anxiety and depression) in non-psychiatric patients treated at hospital clinics. It consists of 14 items with 7 items relating to anxiety and to depression respectively. Each item is scored from 0 to 3 therefore scores for each subscale range from 0 to 21 with higher scores indicating higher levels of anxiety and depression. The scores were categorized as follows: 0 to 7 was normal, 8 to 10 was suggestive, and 11 to 21 was case.
Time Frame: Baseline and Visit 3 [Month 6]
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Adalimumab
Number analyzed (Participants) | 59
participants
  Normal to Normal | 33
  Normal to Suggestive | 5
  Normal to Case | 2
  Suggestive to Normal | 5
  Suggestive to Suggestive | 7
  Suggestive to Case | 0
  Case to Normal | 1
  Case to Suggestive | 2
  Case to Case | 4

4. Primary Outcome: Change in Hospital Anxiety and Depression Score (HADS) - Depression, From Baseline to After 6 Months of Treatment With Adalimumab
Description: as for outcome 3
Time Frame: Baseline and Visit 3 [Month 6]
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Adalimumab
Number analyzed (Participants) | 59
participants
  Normal to Normal | 47
  Normal to Suggestive | 8
  Normal to Case | 0
  Suggestive to Normal | 0
  Suggestive to Suggestive | 2
  Suggestive to Case | 0
  Case to Normal | 1
  Case to Suggestive | 1
  Case to Case | 0

5. Secondary Outcome: Short Inflammatory Bowel Disease Questionnaire (sIBDQ) Scores by Visit
Description: The sIBDQ is a disease-specific health-related quality of life (HRQoL) questionnaire, able to detect and define meaningful clinical changes in inflammatory bowel disease (IBD) patients by measuring physical, social and emotional status. The sIBDQ consists of 10 questions, each question is scored on a scale from 1 (poor QoL) to 7 (good QoL). The scores are summed up and divided by 10 for a mean score ranging from 1 (poor QoL) to 7 (good QoL). A higher score indicates a better HRQoL.
Time Frame: Visit 1 [Baseline], Visit 2 [Month 3], and Visit 3 [Month 6]
Population: All data were analyzed as observed and missing values were not replaced by any imputation method.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Adalimumab
Number analyzed (Participants) | 77
scores on a scale
  Visit 1 [N=77] | 4.58 (1.21)
  Visit 2 [N=48] | 5.19 (1.01)
  Visit 3 [N=63] | 5.22 (1.06)

6. Secondary Outcome: Harvey-Bradshaw Index (HBI) Scores by Visit
Description: Harvey-Bradshaw Index (HBI) is for use in the assessment and quantification of symptoms and the present level of disease activity of patients with Crohn's disease. It is a validated clinical index for Crohn's disease, including the 5 categories of: general well-being, abdominal pain, number of liquid stools, abdominal mass and complications. The score ranges from 0 to 25 with higher scores indicating higher disease activity. The scores were classified as follows: less than 5 is remission, 5 to 7 is mild, 8 to 16 is moderate, and greater than 16 is severe.
Time Frame: Visit 1 [Baseline], Visit 2 [Month 3], and Visit 3 [Month 6]
Population: All data were analyzed as observed and missing values were not replaced by any imputation method.
Measure: Number; unit: participants
Arm/Group | Adalimumab
Number analyzed (Participants) | 76
participants
  Visit 1: Remission [N=76] | 22
  Visit 1: Mild [N=76] | 26
  Visit 1: Moderate [N=76] | 27
  Visit 1: Severe [N=76] | 1
  Visit 2: Remission [N=50] | 38
  Visit 2: Mild [N=50] | 6
  Visit 2: Moderate [N=50] | 6
  Visit 2: Severe [N=50] | 0
  Visit 3: Remission [N=60] | 39
  Visit 3: Mild [N=60] | 11
  Visit 3: Moderate [N=60] | 10
  Visit 3: Severe [N=60] | 0

7. Secondary Outcome: State Trait Anxiety Index (STAI) State Scores by Visit
Description: as for outcome 1
Time Frame: Visit 1 [Baseline], Visit 2 [Month 3], and Visit 3 [Month 6]
Population: All data were analyzed as observed and missing values were not replaced by any imputation method.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Adalimumab
Number analyzed (Participants) | 79
scores on a scale
  Visit 1 [N=79] | 40.4 (10.7)
  Visit 2 [N=49] | 38.1 (10.2)
  Visit 3 [N=61] | 38.0 (10.5)

8. Secondary Outcome: State Trait Anxiety Index (STAI) Trait Scores by Visit
Description: as for outcome 1
Time Frame: Visit 1 [Baseline], Visit 2 [Month 3], and Visit 3 [Month 6]
Population: All data were analyzed as observed and missing values were not replaced by any imputation method.
Measure: Mean (Standard Deviation); unit: scores on a scale
Groups:
- Adalimumab: 40 mg every other week via subcutaneous injection according to Summary of Product Characteristics (SmPC)
Arm/Group | Adalimumab
Number analyzed (Participants) | 77
scores on a scale
  Visit 1 [N=77] | 38.9 (10.8)
  Visit 2 [N=48] | 38.1 (11.2)
  Visit 3 [N=61] | 37.0 (9.5)

9. Secondary Outcome: Hospital Anxiety and Depression Score (HADS) - Anxiety Scores by Visit
Description: as for outcome 3
Time Frame: Visit 1 [Baseline], Visit 2 [Month 3], and Visit 3 [Month 6]
Population: All data were analyzed as observed and missing values were not replaced by any imputation method.
Measure: Number; unit: participants
Arm/Group | Adalimumab
Number analyzed (Participants) | 79
participants
  Visit 1: Normal [N=79] | 52
  Visit 1: Suggestive [N=79] | 16
  Visit 1: Case [N=79] | 11
  Visit 2: Normal [N=50] | 32
  Visit 2: Suggestive [N=50] | 12
  Visit 2: Case [N=50] | 6
  Visit 3: Normal [N=61] | 40
  Visit 3: Suggestive [N=61] | 14
  Visit 3: Case [N=61] | 7

10. Secondary Outcome: Hospital Anxiety and Depression Score (HADS) - Depression Scores by Visit
Description: as for outcome 3
Time Frame: Visit 1 [Baseline], Visit 2 [Month 3], and Visit 3 [Month 6]
Population: All data were analyzed as observed and missing values were not replaced by any imputation method.
Measure: Number; unit: participants
Arm/Group | Adalimumab
Number analyzed (Participants) | 79
participants
  Visit 1: Normal [N=79] | 69
  Visit 1: Suggestive [N=79] | 5
  Visit 1: Case [N=79] | 5
  Visit 2: Normal [N=50] | 41
  Visit 2: Suggestive [N=50] | 7
  Visit 2: Case [N=50] | 2
  Visit 3: Normal [N=61] | 49
  Visit 3: Suggestive [N=61] | 11
  Visit 3: Case [N=61] | 1

ADVERSE EVENTS:
Time Frame: From the time of informed consent up to 70 days following the intake of the last dose of physician-prescribed treatment
Description: Only Serious Adverse Events were required to collect, therefore other Adverse Events were not collected
Arm/Group | Adalimumab
Serious Adverse Events (participants affected / at risk) | 9/83
Other Adverse Events (participants affected / at risk) | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Adalimumab (N=83)
Back pain (Musculoskeletal and connective tissue disorders) | 1
Hyperemesis gravidarum (Pregnancy, puerperium and perinatal conditions) | 1
Drug eruption (Skin and subcutaneous tissue disorders) | 1
Bone lesion (Musculoskeletal and connective tissue disorders) | 1
Drug ineffective (General disorders) | 1
Paraesthesia (Nervous system disorders) | 1
Anal Abscess (Gastrointestinal disorders) | 2
Crohn's disease (Gastrointestinal disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.